CLINICAL TRIAL: NCT00860197
Title: Effect of Coffee Consumption on Immune and Inflammatory Status in Elderly
Brief Title: Immune Benefits of Coffee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Daniel Bunout, MD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: immunecoffee
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Immune Senescence; Low-grade Inflammation
Keywords: Coffee; Elderly; Immune response; Inflammatory status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No coffee
- Group 1 (Experimental): Fully torrefied coffee
  Interventions: Dietary Supplement: Fully torrefied coffee
- Group 2 (Experimental): Partially torrefied coffee
  Interventions: Dietary Supplement: Partially torrefied coffee

INTERVENTIONS:
Dietary Supplement: Fully torrefied coffee — Fully torrefied coffee
  Arms: Group 1
Dietary Supplement: Partially torrefied coffee — Partially torrefied coffee
  Arms: Group 2

SUMMARY:
This study will assess whether coffee consumption:

* increases immune responses
* decreases inflammatory status

DETAILED DESCRIPTION:
Epidemiological studies suggest that coffee consumption is associated with protective effects against several types of chronic diseases. Recent data have shown that certain coffee components may possess anti-inflammatory and immune-enhancing properties. Low-grade inflammation and poor capacity of immune response is highly prevalent in elderly subjects.

The purpose of this study is to evaluate whether coffee consumption improves immune and inflammatory status in healthy elderly subjects. To sort out the role of antioxidants, we will test 2 different soluble coffee, i.e. fully torrefied coffee and partially torrefied coffee.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, self-sufficient, free-living Chilean elderly
* Having the ability to comprehend the procedures of the study
* Having obtained his/her informed consent after verbal and written information

Exclusion Criteria:

* Subjects drinking more than 2 cups of coffee per day
* Subjects with rapidly deteriorating health status at enrolment in the study
* Subjects with terminal or acute disease, or unstable health status
* Subjects with chronic disease: chronic respiratory illness; chronic diseases of the pulmonary or cardiovascular systems (including asthma); chronic metabolic disease (diabetes); chronic renal disease, organ failure
* Subjects with serious neurological disorder, including dementia (MMSE < 20) or Alzheimer's disease
* Subjects who have experienced rapid weight loss, chronic diarrhea (loose stools, 3 times daily), or Crohn's (IBD)
* Subjects with gastrointestinal problems
* Subjects with a hospitalization planned during this study
* Subjects who have received any antibiotic treatment during the last 3 months prior to the beginning of this study
* Subjects who had a colonoscopy performed during the last 3 months prior to the beginning of this study
* Subjects with immune deficiency diseases (e.g. HIV infection)
* Subjects with a history of allergy - especially to egg protein, egg, shellfish or the antibiotics polymyxin or neomycin
* Subjects receiving medication that may influence the immune system (i.e. corticosteroids, immuno-suppressors and immuno-modulators, antimicrobials)
* Subjects who have received any vaccination during the last 15 days prior to baseline
* Subjects who are expected to be non-compliant
* Subjects currently participating or having participated in another clinical trial during the last 3 months prior to the beginning of this study
* Subjects participating in another research study involving any type of medication related to the study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
NK-cell activity | will be measured before and after 30 days +/- treatment
Tuberculin test | will be measured before and after 30 days +/- treatment
Inflammatory status | will be measured before and after 30 days +/- treatment

SECONDARY OUTCOMES:
Gut microbiota profiling | will be measured before and after 30 days +/- treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bunout, MD, Principal Investigator — INTA University of Chile, Santiago, Metropolitana, Chile
Locations (1):
- INTA University of Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- See also: Web site of INTA University of Chile — http://www.inta.cl